CLINICAL TRIAL: NCT02265562
Title: Evaluation of the Effect of Rectal Misoprostol on Blood Loss During Abdominal Hysterectomy: A Double Blind Randomized Controlled Trial.
Brief Title: Rectal Misoprostol and Blood Loss During Abdominal Hysterectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Assistant Professor of Obstetrics & Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10102014
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Blood Loss
Keywords: Hysterectomy; Misoprostol; Blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): 60 minutes before the surgery 400 μg of misoprostol (2 tablets of 200 μg) inserted rectally
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): 60 minutes before the surgery 2 tablets of placebo tablets inserted rectally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 60 minutes before the surgery 400 μg of misoprostol (2 tablets of 200 μg) inserted rectally
  Other Names: prostaglandin E1 analogue
  Arms: Misoprostol
Drug: Placebo — 60 minutes before the surgery 2 tablet of placebo inserted rectally
  Other Names: Dizirest B6
  Arms: Placebo

SUMMARY:
Hysterectomy, as any major operation, can cause complications, as hemorrhage which may occur in some cases and sometimes requiring blood transfusion. Recent study proved that misoprostol success in reducing blood loss during total abdominal hysterectomy when used once before the surgery.

DETAILED DESCRIPTION:
In this study we tried to assess the efficacy of misoprostol in minimize blood loss during hysterectomy when used as single preoperative dose via rectal route. The reduction of blood flow may be due to the combined effect of myometrial contraction and vasoconstrictive effect

ELIGIBILITY:
Inclusion Criteria:

A- Age: adult female >18 years old. B- Any women undergoing abdominal hysterectomy. C- No contraindications to misoprostol.

Exclusion Criteria:

A -Women with any contraindications to misoprostol including heart disease, mitral stenosis , severe hypertension ( diastolic pressure over100mm Hg) , hematologic disorders (as sickle cell anemia ), glaucoma, bronchial asthma, liver disease.

B- Known history of or active medical disorder as DM . C- Pelvic endometriosis and adnexal mass. D- Those who had undergone previous myomectomy. E- Women who received GnRH analogues and mifepristone and who are allergic to prostaglandins.

F- Women with mental impairment or incompetent in giving consent. G- Women who don't wish to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 8 months
  amount of intra-operative blood loss

SECONDARY OUTCOMES:
postoperative hemoglobin level | 8 months
  level of serum hemoglobin postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-khyatat, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo University hospiatl, Cairo, Egypt